CLINICAL TRIAL: NCT03304535
Title: The Impact of a Social Worker in a Glaucoma Eye-Care Service: A Prospective Study
Brief Title: Social Worker in an Eye-Care Service
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Scott Fudemberg, MD, Principal Investigator, Wills Eye
Other Study IDs: IRB#15-XXX
Record Dates: First submitted 2016-02-22; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Glaucoma
Keywords: Glaucoma; Social Worker
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to determine whether involvement with a social worker helps reduce distress, depression, and increase patient activation in participants over a 6 month intervention period. The study will also describe common barriers to care that participants face.

DETAILED DESCRIPTION:
An appointment will be scheduled for participant to meet with a social worker. The appointment may happen on day of participant's scheduled clinic appointment or on another mutually decided upon date and time. Should participant choose to participate, this first visit will be Visit 1 for the study.

Visit 1: Baseline

Informed consent will be obtained demonstrating an interest in participating.

A visit with the social worker will take place during Visit 1. This session will be held in a private office and allows participant time for discussion regarding any challenges, struggles and/or barriers they may be experiencing.

The following baseline questionnaires/surveys will be administered:

Modified Patient Activation Measure - measures participant confidence in taking care of their own health.

Distress Thermometer - measures participant distress level during the past week.

Patient Health Questionnaire -measures depression symptoms and severity if any.

Clinical information will be taken from participant's medical record. There may be follow-up questions related to data if information is unclear or incomplete.

Upon completion of Visit 1, participant will receive a satisfaction survey to evaluate how participant satisfaction with social worker interaction.

Social Worker Interventions: After Visit 1 and before Visit 2

The social worker will develop an intervention for participant during Visit 1 appointment. As many calls or in person meetings participant requires will take place. There will be no limit and it will be determined by participant's needs.

Visit 2: Follow-up After 6 Months

Upon completion of participant's six month follow-up in the study, the following questionnaires/surveys will be administered:

Modified Patient Activation Measure - measures how confident participant is at taking care of their own health.

Distress Thermometer - measures how much distress participant has been experiencing in the past week.

Patient Health Questionnaire - measures if participant has symptoms of depression and the severity of those symptoms.

Satisfaction Survey - measures how satisfied participant is with the social worker interaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at Wills Eye Hospital in the Glaucoma Service
* Glaucoma of any type, characterized by glaucomatous optic neuropathy and corresponding visual field (VF) defect
* Referred to staff social worker for intervention
* Ability to read, write, speak and understand English

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with any type of Glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in response to Patient Health Questionnaire 9 | 6 months
  Measures participant levels of depression based on questions related to depressive symptoms. The investigator will assess change in the number of participants with major, moderate, and minimal depressive symptoms.

SECONDARY OUTCOMES:
Change in response to Distress thermometer | 6 months
  Measures participant level of distress on a scale of 1 to 10 and asks additional questions regarding contributors to distress.
Change in response to Modified Patient Activation Measure 13 | 6 months
  Measures participant self-capacity for and confidence regarding glaucoma management.
Descriptive results of the Social Worker Baseline Assessment | 6 months
  Social worker will assess each participant's internal and external barriers to care, limitations, and strengths that may help them to manage their glaucoma.

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Fudemberg, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fudemberg SJ, Amarasekera DC, Silverstein MH, Linder KM, Heffner P, Hark LA, Waisbourd M. Overcoming Barriers to Eye Care: Patient Response to a Medical Social Worker in a Glaucoma Service. J Community Health. 2016 Aug;41(4):845-9. doi: 10.1007/s10900-016-0162-1. PMID 26860278